CLINICAL TRIAL: NCT02025270
Title: Using of Bone Marrow Derived Mesenchymal Stem Cells For Treatment of Azoospermic Patients
Brief Title: MSCs For Treatment of Azoospermic Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Sayed Bakry, Associate Professor , Consultant of Separation and Culturing of Stem Cells, Al-Azhar University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: AZH010066099; Azhar23052011 (Other Grant/Funding Number: Al Azhar University)
Record Dates: First submitted 2013-12-13; First posted 2014-01-01 (Estimated); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Male Infertility
Keywords: Azoospermia, Spermatogonial Arrest, Maturation Arrest.
MeSH Terms: conditions — Infertility, Male; Azoospermia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Laboratory and Clinical (Other): 60 ml of Bone marrow will aspirated for stem cells isolation and preparation. 5 ml of stem cells prepared according to GMP rules injected into rete testis.
  Interventions: Biological: Stem Cells

INTERVENTIONS:
Biological: Stem Cells — 60 ml of bone marrow will aspirated and used for stem cells isolation. Then stem cells will cultured using autologous serum, characterized and prepared using GMP rules and finally injected into rete testis.
  Other Names: Stem Cell Dose; 3-5 Million Autologous MSCs Injected into rete testis.

SUMMARY:
In this study, we performed autologous BMDMSC transplantation to the testis of Azoospermic patients in a trial to enhance and activate the spermatogonial stem cells of the testis and aiming to produce motile sperm.

DETAILED DESCRIPTION:
Bone marrow aspirated and stem cells were isolated, cultured and characterized using flow cytometer. Stem cells prepared according to GMP regulations then injected into rete testis using special syringe. Patients follow up will carried out for a year , three month interval. FSH, testosterone, testicular size as well as sexual potency will assessed every three months.

ELIGIBILITY:
Inclusion Criteria:

* All Non obstructive Azoospermic Patients.
* Azoospermic Patients due to Administration of Chemo/Radiotherapy.

Exclusion Criteria:

* Patients with Testicular Cancer.
* Patients with Complete Deletion of Chromosome Y AZF (a,b,c) Regions.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-10-15 (Actual); Primary Completion 2016-10-15 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
All Cases Improvement | One Year (12-Month)
  Hormonal Assessment: Serum (Testosterone , FSH, LH and Prolactin). Testicular Size. Sexual Potency.

SECONDARY OUTCOMES:
All Cases Fertility Improvement | One Year (12-Month)
  Hormonal Assessment: Serum (Testosterone , FSH, LH and Prolactin) Testicular size and Sexual Potency.

CONTACTS AND LOCATIONS:
Overall Officials: Taimour M Khalifa, MD Professor, Principal Investigator — Al-Azhar University; Sayed Bakry, PhD, Study Director — Al-Azhar University; Saad Moneer, MSc, Study Chair — Al-Azhar University; Ahmed Kadeh, MSc, Study Chair — Al-Azhar University
Locations (1):
- Al Azhar University , School of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes